CLINICAL TRIAL: NCT02154802
Title: Increasing HIV Testing in Urban Emergency Departments Via Mobile Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Ian Aronson, Principal Investigator, National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 1R34DA037129-01A1 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: HIV Testing

ARMS (4):
- video: community member (Experimental): Participant watches video of a community member
  Interventions: Behavioral: video: community member
- video: physician (Experimental): Participant watches video of a physician
  Interventions: Behavioral: video: physician
- video: choice of video (Experimental): Participant can choose to watch video of either the community member of the physician
  Interventions: Behavioral: video: choice of video
- no video (No Intervention)

INTERVENTIONS:
Behavioral: video: community member
  Arms: video: community member
Behavioral: video: physician
  Arms: video: physician
Behavioral: video: choice of video
  Arms: video: choice of video

SUMMARY:
Because people with undiagnosed HIV will not receive treatment and may unknowingly infect others, the investigators propose a mobile computer-based video intervention to increase HIV test rates in high volume urban hospital emergency departments (EDs). EDs offer important points of contact for many of those at greatest risk for HIV. Unfortunately, when ED patients are offered routine HIV testing, most decline. Our proposed intervention builds upon initial findings from a trial our research team conducted with patients who declined HIV testing. The intervention, grounded in the Information-Motivation and Behavioral Skills model (IMB), showed an onscreen physician explaining the importance of HIV testing (to build knowledge and motivation) and modeling a rapid HIV test (to increase motivation and behavioral skill). This brief intervention had a potent effect: a third accepted HIV testing post-intervention. While this preliminary study is highly encouraging, it revealed a number of other critical research questions. First, it remains unclear what intervention component most strongly contributed to patients' decisions to test: the video content or the offer of an HIV test by a computer rather than a person. Second, consistent with the literature, participants indicated a community member disclosing positive HIV status onscreen would increase the proportion of patients who test. Third, results suggest there is individual variation in the extent to which behavior is more strongly influenced by onscreen community members or experts (e.g. physicians). Therefore, the goal of the present study, guided by the IMB model, is to determine how the investigators can refine mobile computer-based interventions to maximize HIV testing rates among patients who initially decline to test in the ED. At the end of the computerized intervention, onscreen text will ask patients if they would agree to an HIV test. Those who agree will be tested by ED staff. The study's endpoint will be post-intervention HIV test rates. The investigators' study will inform scalable interventions for underserved populations nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Capable of providing informed consent
* Reads English
* Declined HIV test offered by hospital staf at triage

Exclusion Criteria:

* intoxicated
* a prisoner
* known to be HIV positive
* presenting to the hospital for a psychiatric problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who accept an HIV test after completing the intervention | Day 1
  The intervention computers will show participants a set of videos and data collection instruments. When the participant has watched the video and responded to all instruments, the computers will ask patients if they would like an HIV test. Answers are yes or no.

SECONDARY OUTCOMES:
Knowledge change | Baseline, Day 1
  The intervention computers will display a set of HIV-related knowledge questions before and after a video segment. This will enable the investigators to examine potential increases in participants' knowledge after watching a video.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Emergency Department, New York, New York, United States